CLINICAL TRIAL: NCT04613297
Title: HLA-G Immuno-Inhibitor Checkpoint Study in Patients With COVID-19 Infection: Molecular and Cellular Assessment
Acronym: HLA-G-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020_0082
Record Dates: First submitted 2020-11-02; First posted 2020-11-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Covid19
Keywords: HLA-G
MeSH Terms: conditions — COVID-19 | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COVID-19 uninfected patients (Other): Patient with negative PCR result
  Interventions: Other: Baseline blood sample
- non-hospitalized COVID-19 infected patients (Other): Patient with positive PCR result who does not require hospitalization for COVID-19
  Interventions: Other: Baseline blood sample
- hospitalized COVID-19 infected patients (Other): Patient with positive PCR who require hospitalization for COVID-19
  Interventions: Other: Baseline and during hospitalization blood samples

INTERVENTIONS:
Other: Baseline and during hospitalization blood samples — Blood sample will be performed at the inclusion visit for all patient and for the hospitalized COVID-19 infected patients, extra-blood samples will be performed :
  * at day 3
  * day 5 and
  * In case of aggravation
  * At the discharge from hospital
  Arms: hospitalized COVID-19 infected patients
Other: Baseline blood sample — Blood sample will be performed at the inclusion visit only
  Arms: COVID-19 uninfected patients; non-hospitalized COVID-19 infected patients

SUMMARY:
The aim of the research is to study the immune checkpoint linked to the HLA-G molecule in the dysregulation of the control of COVID-19 infection.

DETAILED DESCRIPTION:
Single-center, prospective, open-ended, interventional study with minimal risks and constraints. Patients will be divided into 3 groups: patients not infected with COVID-19, patients infected with COVID-19 not hospitalized, patients infected with COVID-19 hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Patient with possible or confirmed infection by COVID-19

Exclusion Criteria:

* Patient without liberty or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Comparison of the percentage of T cells expressing the HLA-G receptor ILT2 (CD3+CD4+ILT2+ T cells, and CD3+CD8+ILT2+ T cells) between the 3 groups of patients. | 1 month
  The CD3 + T lymphocyte cell populations (CD4 + ILT2 + and CD8 + ILT2 +) will be compared between the groups of patients
Comparison of the expression of circulating soluble HLA-G, between the groups of patients. | 1 day
  Blood levels of soluble HLA-G and plasma microvesicles with expression of HLA-G will be compared between the groups of patients.

SECONDARY OUTCOMES:
1 month survival | 1 month
  Vital status collected 1 month post inclusion for all the patients
Assessment of the severity of the disease according to the isoform of HLA-G | 1 month
  Comparison of the isoforms (alleles) of HLA-G regarding the severity of the disease for the infected patients.
Comparison of the expression of one of the cell receptors of the SARS-CoV-2 virus, called BSG (Basigin), whose expression is modified by the interaction between HLA-G. | 1 day
  The expression of the BSG cell receptor induced by HLA-G will be compared between COVID19 patients and uninfected patients.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BRUGIERE, PhD, Principal Investigator — Hopital Foch
Locations (1):
- Foch hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: No